CLINICAL TRIAL: NCT04261881
Title: Nutraceutical Support of Fatigue Reduction, Improved Physical, Mental and Cognitive Function and Improved Mitochondrial Function
Brief Title: Nutraceutical Support of Fatigue Reduction, Improved Physical, Mental & Cognitive Function and Mitochondrial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NIS143-004
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-02

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutraceutical intervention, 5 capsules twice daily. (Active Comparator): Participants will consume the nutraceutical blend ATP-Fuel at 5 capsules twice daily.
  Interventions: Dietary Supplement: ATP-Fuel
- Nutraceutical intervention, 3 capsules once daily. (Active Comparator): Participants will consume the nutraceutical blend ATP-II at 3 capsules once daily.
  Interventions: Dietary Supplement: ATP-II
- Nutraceutical intervention, 3 capsules twice daily. (Active Comparator): Participants will consume the nutraceutical blend ATP-II at 3 capsules twice daily.
  Interventions: Dietary Supplement: ATP-II

INTERVENTIONS:
Dietary Supplement: ATP-Fuel — 5 capsules daily with breakfast and 5 capsules daily with lunch
  Arms: Nutraceutical intervention, 5 capsules twice daily.
Dietary Supplement: ATP-II — 3 capsules daily with breakfast
  Arms: Nutraceutical intervention, 3 capsules once daily.
Dietary Supplement: ATP-II — 3 capsules daily with breakfast and 3 capsules daily with lunch
  Arms: Nutraceutical intervention, 3 capsules twice daily.

SUMMARY:
The purpose for this protocol is to perform an open-label human clinical pilot study on the effects of consumption of two nutraceutical blends in subjects with long-term unexplained fatigue interfering with daily living.

DETAILED DESCRIPTION:
This is an open-label human clinical study to evaluate the effects of consumption of the nutraceutical product ATP-Fuel, compared to the nutraceutical product ATP-II. The study participants will be randomized to one of three groups: consuming ATP-Fuel (5 capsules, twice daily); consuming ATP-II (3 capsules, once daily); or consuming ATP-II (3 capsules, twice daily). The study is of 8 weeks' duration, with evaluation at baseline, 1, 4, and 8 weeks of product consumption.

At each visit the following measurements and procedures are performed: Blood pressure, questionnaires pertaining to fatigue, pain and wellness, and a blood draw. The blood is used for testing of lipid peroxidation and mitochondrial volume and metabolic activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult people of either gender;
* Age 18-75 years (inclusive);
* BMI between 18.0 and 34.9 (inclusive);
* Experiencing fatigue, at a level that moderately to severely interferes with daily activities, for the past 6 months.

Exclusion Criteria:

* Cancer during past 12 months;
* Chemotherapy during past 12 months;
* Currently taking blood thinning medication (81mg aspirin allowed);
* Getting regular joint injections (such as cortisone shots);
* Have received a cortisone shot within past 12 weeks;
* Major surgery within the past 3 months;
* Major trauma within the past 3 months;
* Any other significant disease or disorder that the investigator judges may put the subject at risk because of participation in the study, or may influence the result of the study;
* Known food allergies or sensitivities related to the test products;
* Participation in another research study involving an investigational product in the past month;
* Planned surgery within 2 weeks of completing the study;
* Previous major surgery to stomach or intestines [(absorption of test product may be altered) minor surgery is not a problem, including appendix and gallbladder removal];
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Women who are pregnant, nursing, or trying to become pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Change in fatigue level from baseline | 8 weeks
  Piper Fatigue Scale - Change from baseline will be evaluated. Each question scores 0-10, 22 questions.

SECONDARY OUTCOMES:
Change in primary and secondary pain levels from baseline | 8 weeks
  Pain questionnaire: Scale 0-10, with 0 being pain-free and 10 being the most pain. Change from baseline will be evaluated.

OTHER OUTCOMES:
Change in physical and mental energy, cognitive function and general wellness from baseline | 8 weeks
  Thirty-point questionnaire. Each question scores 0-10, max score therefore 300. Change from baseline will be evaluated.
Change in mitochondrial mass and mitochondrial membrane potential from baseline | 8 weeks
  Mean fluorescence
Change in lipid peroxidation from baseline | 8 weeks
  Malondialdehyde level µg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Jensen, PhD, Principal Investigator — NIS Labs
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

REFERENCES:
- [Derived] Hamilton D, Jensen GS. Nutraceutical Support of Mitochondrial Function Associated With Reduction of Long-term Fatigue and Inflammation. Altern Ther Health Med. 2021 May;27(3):8-18. PMID 33882028